CLINICAL TRIAL: NCT03232177
Title: A Multicenter, Open-label, Clinical Study for Efficacy and Safety Evaluation of Anagrelide in Patients With Treatment-naïve, High-risk Essential Thrombocythemia as a Primary Treatment
Brief Title: Anagre Cap. in Patients With High-Risk Essential Thrombocythemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YMC018
Record Dates: First submitted 2017-07-11; First posted 2017-07-27 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Essential Thrombocythemia
MeSH Terms: conditions — Thrombocythemia, Essential

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anagre Cap. (Experimental): twice a day
  Interventions: Drug: Anagre Cap.

INTERVENTIONS:
Drug: Anagre Cap. — from 0.5mg twice a day to maximally increase total10mg in 8 weeks and maintain maximal tolerable dose to 104 weeks

SUMMARY:
This study is to evaluate the efficacy and safety according to incremental dosing for 8 weeks and duration of administration for 1 year in patients with high-risk essential thrombocythemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with essential thrombocythemia according to WHO 2008
* Any of the following as high-risk patient

  * Over 60 years old
  * >100 X 10^4/ul of platelet count
  * increased more than 300K of platelet count in 3 months
  * Hypertension, diabetes, past history of thromboembolic bleeding

Exclusion Criteria:

* Patients with an adverse drug reaction or intolerability to anagrelide
* Any of the following cardiac abnormalities;

  * Complete left bundle branch block on ECG
  * Patients using a pacemaker
  * Patients with a family history of congenital QT prolongation syndrome or known QT prolongation syndrome
  * Currently, there is no clinically uncontrolled ventricular or atrial tachycardia
  * Clinically significant bradycardia (<less than 50 per minute)
  * History of clinically proven myocardial infarction and unstable angina within 3 months
* Pregnant women, nursing mothers

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2020-12-05 (Actual); Study Completion 2020-12-05 (Actual)

PRIMARY OUTCOMES:
response rate for less than 60 X 10^4/ul in platelet count | at week 8

SECONDARY OUTCOMES:
response rate for less than 60 X 10^4/ul in platelet count | at week 52
changes from baseline in 50% reduction rate in platelet count | up to 52 weeks
response rate for less than 40 X 10^4/ul in platelet count | up to 52 weeks
cumulative incidence of essential thrombocythemia related events (e.g thromboembolic or hemorrhagic events) | at 52 week
incidence of adverse events | up to 52 weeks

OTHER OUTCOMES:
expression of MPN-oncogene(JAK2/CALR/MPL) | at 52 week
  association of known MPN-oncogene(JAK2/CALR/MPL) with epigenetic modifiers, mRNA splicing, oncogene and other minor somatic mutations
genomic biomarker search for prediction of side effects of anagrelide | at 52 week

CONTACTS AND LOCATIONS:
Locations (21):
- South Korea (21):
  - National Health Insurance Service Ilsan Hospital, Goyang-si, Gyeonggi-do
  - The Catholic University of Korea. ST. Vincents Hospital, Suwon, Gyeonggi-do
  - Hallym UNIV. Medical Center, Anyang
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook national university hospital, Daegu
  - Dongguk University Medical Center, Goyang
  - Cheonnam National University Hwasun Hospital, Hwasun
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Jeju National University Hospital, Jeju City
  - Pusan National University Hospital, Pusan
  - Ewha Wonans University Mokdong Hospital, Seoul
  - Hallym UNIV. Medical Center, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - SMG - SNU Boramae Medical Center, Seoul
  - Soon Chun Hyang University Hospital Seoul, Seoul
  - Veterans Health Service medical Center, Seoul
  - Yonsei University Health System, SEVERANCE HOSPITAL, Seoul

IPD SHARING:
Plan to Share IPD: No